CLINICAL TRIAL: NCT06388213
Title: Investigation of Gastric Emptying in Patients Treated With GLP-1 Receptor Agonists
Brief Title: Investigation of the Evolution of Gastric Emptying by Gastric Ultra Sonography in Patients Treated With GLP-1 Receptor Agonists on a 7 Days Pausing Period.
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Eduardo Schiffer, Professor, University Hospital, Geneva
Other Study IDs: GLP-1 RA patients GE by GUS
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2; Anesthesia; Pulmonary Aspiration of Gastric Contents
Keywords: Glucagon Like Peptide 1 Receptors Agonists; Gastric Emptying; Gastric Ultrasound
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Non GLP-1 RA group: Patient aged 18 years or older in healthy condition with no gastroparetic treatment and without history of gastro-intestinal pathology, respecting fasting period of 6 hours for solid or thick liquid (juice, milk, sparkling water and soda) and 2 hours for clear liquid (still water, black coffee or tea).
  Interventions: Device: Gastric Ultrasonography
- GLP-1 RA group: Patients aged 18 years or older, treated with GLP-1 receptor agonists, respecting fasting period of 6 hours for solid or thick liquid (juice, milk, sparkling water and soda) and 2 hours for clear liquid (still water, black coffee or tea).
  Interventions: Device: Gastric Ultrasonography

INTERVENTIONS:
Device: Gastric Ultrasonography — Evaluation of cross sectional area of the antrum by gastric ultrasonography in healthy patients and in patient treated by GLP-1 receptor agonists after a fasting period (6 hours for solid and 2 hours for clear liquids). For the GLP-1 receptor agonists group the gastric ultrasonochography will be repeated each 2 days during 7 days. In the non GLP-1 receptors agonists group the evaluation will be executed one time.

SUMMARY:
Glucagon-like-peptide-1 is a hormone released by the gut enteroendocrine cells. Its secretion occurs after each meal to enable production of insulin and inhibits the production of glucagon to lower after meal glycemia. It also inhibits gastric emptying and food intake. GLP-1 RA plays a role on GLP-1 receptors present on islet beta cells and delta cells of the pancreas to control insulin. GLP-1 receptors are also present in multiple region of the central nervous system such as the hypothalamus and hindbrain where it results in reducing food intake. For anesthesiologist it is important to understand how GLP-1 RA influence gastric emptying. Indeed, respecting a fasting period (6 hours for solid and 2 hours for liquid) before each surgery is one of the cornerstones of anesthesiology to significantly reduce the risk of pulmonary aspiration. One of the side effects of GLP-1 RA is slowing gastric emptying and increasing the risk of regurgitation in patient that observed a recommended fasting period. During 2023 a lot of cases reports have emerged of pulmonary aspiration or the presence of a full stomach in patient treated by GLP-1 RA for a type 2 diabetes. Despite recommendations made by the American Society of Anesthesiology, it is still unkown what is the best fasting period and how long patients should pause a long acting GLP-1 RA before surgery. In this observational study, we would like to determine the effect of GLP-1 RA on gastric emptying in patient scheduled for general anesthesia. We will measure and compare residual gastric content with gastric ultrasonography in patients treated by GLP-1 RA and in those who are not. We will also do these comparisons in a group of patients with type 2 diabetes treated by weekly GLP-1 RA at different days after the injection of the medication. Our hypothesis is that we will observe a reduction in gastric residue in patients who stopped weekly GLP-1 RA 7 days prior the examination compared to those who have stopped less days considering the same fasting period. This would lead us to propose an optimal duration of stopping time for GLP-1 inhibitors in the preoperative period.

DETAILED DESCRIPTION:
The study design consists in a prospective monocentric observational study comparing 2 groups of patients either treated by GLP-1 RA (more than 3 months) or without GLP-1 RA treatment. The investigators will perform a gastric echography, in both groups to define gastric residue after a fasting period of at least 6 hours for solids and 2 hours for liquids. Patients will have free access to any eating regimen before fasting. The instructions given to patients will be to stop eating solids 6h and drinking 2h before investigation. Patients will also fill a nutrition booklet which will be analyzed by a nutritionist nurse thereafter. The investigations will be performed at 24h, 48h, 96h and 144h after last injection of GLP-1 RA in the investigation group, and only once in the control group. Gastric echography will be realized using curved ultrasonic probe placed in sagittal plane on the epigastric area under xyphoid appendix and upper to the umbilicus. Visualization of left hepatic lobe, antrum, aorta and upper mesenteric artery will assess good position of the ultrasonic probe. Qualitative observation of antrum will be made to assess antrum volume in recumbent position. A qualitative and quantitative analyze will be performed in right lateral decubitus by measuring atrum cross-sectional area (CSA). Following formula will be used to determine volume of the antrum : Volume (mL) = 27.0 + 14.6 9 x right-lat CSA - 1.28 x age . A full stomach will be considered when solids are observed or if gastric volume is superior to 1,5 ml/kg. An empty stomach is defined when gastric volume is inferior to 1,5 ml/kg. Gastric echography is proceeded by two anesthetists who will be blinded one to the other. CSA will be compared between two investigation groups. Time-course of CSA and presence of solids or liquids will be assessed at all study time-points up to the seventh day in the investigation group. A reduction of 5,5 cm2 of CSA after one week from last injection of GLP-1 RA will be considered significant. Based on a power study it has been evaluated that a sample of 20 patients per group will be necessary to have a power of 80% with an alpha risk of 0,05.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18yrs old treated with GLP-1 receptor agonists for at least three months

Exclusion Criteria:

Patients known for gastrointestinal motility disorders, history of gastric surgery, large hiatal hernia, or inability to lie in the right lateral decubitus position.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with type 2 diabetes treated by an GLP-1 receptors agonists
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change of antral cross sectional area in patients pausing 7 days GLP-1 RA treatment. | 7 days

SECONDARY OUTCOMES:
Time course of change in gastric volume | 7 days

IPD SHARING:
Plan to Share IPD: Undecided